CLINICAL TRIAL: NCT02930889
Title: Prostate Artery Embolization (PAE) for Lower Urinary Tract Symptoms (LUTS) Due to Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAD-2016-24154
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Results first posted 2021-11-15 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-10

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Therapeutic Embolization; Prostatic Artery Embolization
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prostate Artery Embolization (Experimental): Prostate Artery Embolization is a surgical procedure to relieve symptoms of Benign Prostatic Hyperplasia (BPH). Embolizing particles are injected into a target blood vessel to occlude blood flow.
  Interventions: Device: Prostate Artery Embolization

INTERVENTIONS:
Device: Prostate Artery Embolization — Prostate Artery Embolization
  Other Names: PAE

SUMMARY:
This is a investigator-initiated evaluation of the safety and efficacy of treating benign prostatic hyperplasia (BPH) by prostatic artery embolization.

DETAILED DESCRIPTION:
This is a investigator-initiated evaluation of the safety and efficacy of treating benign prostatic hyperplasia (BPH) by prostatic artery embolization.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Male, 45 years or older
* Diagnosis of Lower Urinary Tract Symptoms from Benign Prostatic Hyperplasia refractory to medical therapy for at least 6 months.
* IPSS score at initial evaluation should be greater than 12, and uroflowmetry (Qmax) of <15mL/s (milliliters per second).
* All prostate volumes will be > 40gm
* PSA which meets one of the following criteria:Baseline PSA ≤ 2.5ng/mL, Baseline PSA > 2.5 ng/mL and ≤ 10 ng/mL AND free PSA ≥ 25% of total PSA (no biopsy required);Baseline PSA > 2.5 ng/mL and ≤ 10 ng/mL AND free PSA < 25% of total PSA AND negative prostate biopsy result (minimum of 12 core biopsy) within 12 months;Baseline PSA >10 ng/mL AND negative prostate biopsy result (minimum of 12 core biopsy) within 12 months;Negative prostate biopsy (minimum 12 cores within 12 months) if abnormal digital rectal examination.

Exclusion Criteria:

* Patients with active urinary tract infections or recurrent urinary tract infections (> 2/year), prostatitis, or interstitial cystitis.
* Cases of biopsy proven prostate, bladder, or urethral cancer.
* Patients on long-term narcotic analgesia, androgen therapy, or GNRH (gonadotropin-releasing hormone) analogue therapy who are unwilling to stop therapy for 2 months prior to the study.
* Use of anithistamines, anti-convulsants, and antispasmodics within one week of treatment unless they have been treated with the same drug (at the same dosage) for at least 6 months and has an associated stable voiding pattern.
* Patients who are classified as New York Heart Association Class III (Moderate), or higher, have cardiac arrhythmias, have uncontrolled diabetes, or are known to be immunosuppressed.
* Hypersensitivity reactions to contrast material not manageable with prophylaxis.
* Patients with glomerular filtration rates less than 40 who are not already on dialysis
* Prostate volume <40 mL
* Patients with bilateral internal iliac arterial occlusion
* Patients with causes of bladder obstruction not due to BPH (eg urethral stricture, bladder neck contraction, etc)
* Patients with neurogenic or bladder atonia
* Prior prostatectomy
* Cystolithiasis within the last 3 months
* Patients interested in future fertility
* Patients with a life expectancy less than 1 year
* Patients where embolization is not possible distal to collateral vessels feeding non-prostatic tissue
* Patients with major neurologic illnesses which could have symptoms that may be similar to or confused for BPH (eg Parkinson's disease, multiple sclerosis, Shy-Drager syndrome, spinal cord injury, etc.).
* Patients with urethral stents
* Patients who have undergone prior rectal surgery other than hemorrhoidectomy or pelvic irradiation.
* Patients who have started or changed their dosage of alpha blockers or 5-alpha reductase inhibitors in the month prior to PAE

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jafar Golzarian, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prostate Artery Embolization
Started | 21
Completed | 5
Not Completed | 16
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 6
Not completed — Did not meet inclusion/exclusion criteria | 8

BASELINE CHARACTERISTICS:
Population: All participants from whom data was collected are included.
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events Reported
Description: All adverse events will be collected and reviewed. Adverse events are collected by self-report and medical record. Outcome is reported as the total number of adverse events reported.
Time Frame: 3 Months
Measure: Number; unit: adverse events
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 5
adverse events | 7

2. Primary Outcome: Change in International Prostate Symptom Score
Description: The International Prostate Symptom Score assesses the severity of symptoms in benign prostatic hypertrophy. The questionnaire contains seven items rated on a scale from zero to five. Total scores are a sum of items scores and range from 0 to 35 with higher scores indicating worse BPH symptoms. Outcome is reported as the change in IPS score from baseline to three months.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 5
score on a scale | -15.40 (4.98)

3. Primary Outcome: Change in Quality of Life Scale (QOLS)
Description: Participants will complete the Quality of Life Scale (QOLS), which contains 15 items measuring five domains of quality of life. Total scores are a sum of item scores and range from 16 to 112, with higher scores indicating a better quality of life.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 5
score on a scale | -2.80 (1.30)

4. Primary Outcome: Patient Reported Change in Medication Use
Description: Participants will report change in medication use for prostate symptoms. The number of participants who reduce medications will be reported.
Time Frame: 3 months
Population: Measure was only collected from 2 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 2
Participants | 1

5. Secondary Outcome: Efficacy Measured by Medical Therapy of Prostatic Symptoms Questionnaire or Flow Rate Change
Description: The Medical Therapy of Prostatic Symptoms (MTOPS) Outcome is reported as the number of participants who experience treatment efficacy as defined by an MTOPS composite variable symptom score greater than 30 and/or flow rate change of 15 millimeters per second or greater.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Prostate Artery Embolization
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prostate Artery Embolization (N=5)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prostate Artery Embolization (N=5)
Loose Stool (Gastrointestinal disorders) | 1 (1)
Burning Sensation While Urinating (Renal and urinary disorders) | 1 (2)
Post Procedure Penile Pain (Reproductive system and breast disorders) | 1 (1)
Blood in Urine (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT02930889/Prot_SAP_001.pdf
  • Informed Consent Form (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT02930889/ICF_000.pdf